CLINICAL TRIAL: NCT02032836
Title: A Multi-center, Open-label, Randomized Cross-over Study to Compare the Acute Tolerability and Pharmacokinetics of BAYQ6256 (Iloprost; Ventavis) Inhalation Using the I-Neb Nebulizer and the FOX Nebulizer in Patients With Pulmonary Arterial Hypertension
Brief Title: Comparative PK PD Study in PAH Patients (Fox vs. I-Neb)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 16483; 2013-002783-12 (EudraCT Number)
Record Dates: First submitted 2014-01-09; First posted 2014-01-10 (Estimated); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I-Neb - FOX (Experimental): Part 1: Subjects received single inhalation of 1.25 mcg iloprost using 10 mcg/ml iloprost solution (Ventavis 10) and then 2.5 mcg iloprost using Ventavis 10, both using the FOX nebulizer on Day 1. Part 2: On Day 2, subjects received single inhalation of 5 mcg iloprost using Ventavis 10 with the I-Neb nebulizer; followed by single inhalation of 5 mcg iloprost using 20 mcg/ml iloprost solution (Ventavis 20) with the FOX nebulizer in a cross-over fashion. A washout period of at least 2 hours was maintained between treatments in Part 1 and Part 2. Part 3: Continued on Day 2, and through until Day 30, subjects received multiple inhalations (approximately 6 to 9 inhalations per day) of 5 mcg iloprost using Ventavis 10 with the I-Neb nebulizer for 2 weeks; followed by multiple inhalations (approximately 6 to 9 inhalations per day) of 5 mcg iloprost using Ventavis 20 with the FOX nebulizer for 2 weeks in a cross-over fashion.
  Interventions: Drug: lloprost(Ventavis,BAYQ6252, 20 µg/mL); Drug: lloprost(Ventavis,BAYQ6252, 10 µg/mL)
- FOX - I-Neb (Experimental): Part 1: Subjects received single inhalation of 1.25 mcg iloprost using 10 mcg/ml iloprost solution (Ventavis 10) and then 2.5 mcg iloprost using Ventavis 10, both using the FOX nebulizer on Day 1. Part 2: On Day 2, subjects received single inhalation of 5 mcg iloprost using 20 mcg/ml iloprost solution (Ventavis 20) with the FOX nebulizer; followed by single inhalation of 5 mcg iloprost using Ventavis 10 with the I-Neb nebulizer in a cross-over fashion. A wash-out period of at least 2 hours was maintained between treatments in Part 1 and Part 2. Part 3: Continued on Day 2, and through until Day 30, subjects received multiple inhalations (approximately 6 to 9 inhalations per day) of 5 mcg iloprost using Ventavis 20 with the FOX nebulizer for 2 weeks; followed by multiple inhalations (approximately 6 to 9 inhalations per day) of 5 mcg iloprost using Ventavis 10 with the I-Neb nebulizer for 2 weeks in a cross-over fashion.
  Interventions: Drug: lloprost(Ventavis,BAYQ6252, 20 µg/mL); Drug: lloprost(Ventavis,BAYQ6252, 10 µg/mL)

INTERVENTIONS:
Drug: lloprost(Ventavis,BAYQ6252, 20 µg/mL) — 20 µg/mL iloprost nebulizer solution, inhaled with FOX nebulizer
Drug: lloprost(Ventavis,BAYQ6252, 10 µg/mL) — 10 µg/mL iloprost nebulizer solution, inhaled with I-Neb nebulizer

SUMMARY:
Administration of iloprost aerosol comparing two nebulizers: FOX and I-Neb

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 18 years
* Current diagnosis of pulmonary hypertension (updated Dana Point Classification 1).
* Current inhalative therapy with 5 µg iloprost using the I-Neb nebulizer
* WHO functional class III at the time of the patient's commencement of inhalative therapy with iloprost
* Hemodynamic diagnosis of Pulmonary arterial hypertension(PAH) showing mean pulmonary arterial pressure (mPAP) > 25 mmHg, pulmonary capillary wedge pressure (PCWP) or left ventricular end diastolic pressure (LVEDP) < 15 mmHg and pulmonary vascular resistance (PVR) > 320 dyn•s•cm-5
* If non-specific types of chronic treatment for PAH are being administered: Stable dosage of these for at least the 4 weeks up to screening
* If PAH-specific drug treatments (such as endothelin receptor antagonist (ERA) or phosphodiesterase-5 (PDE5) inhibitors) are being administered: Stable dosage of these for at least the 3 months up to screening.

Exclusion Criteria:

* PAH related to any other etiology, especially to pulmonary veno-occlusive disease (PVOD)
* Clinically relevant obstructive lung disease
* Evidence of thromboembolic disease (probable pulmonary embolism) within 3 years before screening
* Cerebrovascular events within 3 months before screening
* Atrial septostomy within the 6 months before screening
* Severe arrhythmia, or severe coronary heart disease or unstable angina, or myocardial infarction within 6 months before screening, or congenital or acquired valvular defects with clinically relevant myocardial function disorders unrelated to PAH
* Systolic blood pressure < 85 mm Hg, or uncontrolled systemic hypertension (systolic BP > 160 mmHg or diastolic BP > 100 mmHg)
* Hepatic impairment (Child Pugh B, C) or chronic renal insufficiency (creatinine > 2.5 mg/dl) and /or requirement of dialysis
* Clinically relevant bleedings disorders or conditions with increased risk for hemorrhages (active ulcers, trauma etc.)
* Addition or dose change of PAH specific drug treatments such as ERA or PDE5 inhibitors within 3 months before screening, or addition or dose change of non-specific treatments for PAH such as calcium channel blockers, nitrates, digitalis, diuretics within 4 weeks before Screening, or any kind of prostanoid other than those mentioned in inclusion criteria within less than 5 half-lives before treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-03-10 (Actual); Primary Completion 2015-01-07 (Actual); Study Completion 2017-09-29 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with a meaningful maximum increase (i.e. >=25%) in heart rate AND/OR a meaningful maximum decrease (i.e. >=20%) in systolic blood pressure within the 30 minutes after the start of inhalation | multiple measurements within 30 minutes after iloprost inhalation

SECONDARY OUTCOMES:
Maximum change in systolic, diastolic and mean arterial blood pressure | From baseline to multiple BP measurements within 2 hours after iloprost inhalation
Maximum change in heart rate within the 30 minutes following inhalation | From baseline to multiple HR measurements within 30 minutes after iloprost inhalation
Maximum change in oxygen saturation within the 30 minutes following inhalation using finger pulse oxymetry | From baseline to multiple measurements within 30 minutes after iloprost inhalation
AUC (area under the plasma concentration curve of BAYQ6256 from zero to infinity) | Multiple timepoints up to 1 hour
Maximum observed drug concentration in plasma after single dose administration | Multiple blood sampling within 60 minutes after Ventavis inhalation and subsequent iloprost bioanalytics
Time to reach maximum drug observed concentration in plasma after single dose | Multiple blood sampling within 60 minutes after Ventavis inhalation and subsequent iloprost bioanalytics
half-life (associated with terminal slope) | Multiple blood sampling within 60 minutes after Ventavis inhalation and subsequent iloprost bioanalytics

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (6):
- Graz, Styria, Austria
- Germany (5):
  - München, Bavaria
  - Würzburg, Bavaria
  - Giessen, Hesse
  - Cologne, North Rhine-Westphalia
  - Hamburg